CLINICAL TRIAL: NCT01032096
Title: The Neuroendocrine, Metabolic, Inflammatory and Immune Responses to Routine Head and Neck Surgery. An Observational Pilot Study
Brief Title: The Physiological Response to Routine Head and Neck Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Dr Craig Carr, Royal Marsden NHS Foundation Trust
Other Study IDs: CCR3168
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of this pilot study is to observe and document the range of changes in the blood concentrations of certain hormones, inflammatory chemicals and immune chemicals in response to the stimulus of Head and Neck cancer

DETAILED DESCRIPTION:
This project is in keeping with the strategy of the anaesthetic and intensive care departments to push towards greater understanding of the immune, metabolic and inflammatory changes associated with surgery and how these may be modified through use of different anaesthetic and intensive care techniques. Through increased understanding of the stress, inflammatory and immune responses to surgery we may be able to modulate peri-operative care to reduce cytotoxic(Natural Killer and Cytotoxic T cell) immunosuppression and hence micrometastatic spread at the time of surgery in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Elective unilateral neck dissections (Levels I-V) and/or Hemithyroidectomy surgery.
* Royal Marsden Hospital patients with head and neck cancer - all histological sub-types.
* Capable of providing informed consent
* Age >17
* American Society of Anaesthesiologists Classification I-III.

Exclusion Criteria:

* Past history of ipsilateral neck dissection.
* Bilateral neck dissection
* A recent course of systemic steroids (< 3 months)
* Pregnancy
* Involvement in drug trials
* On following medications: Interleukins, Interferons, Immunosuppressants and long term opiates
* Recent Synacthen Test (within 48 hours)
* Emergency surgery
* American Society of Anaesthesiologists Classification IV-V.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of cancer involving the head and neck region of the body.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The maximum increase (from baseline to day 3 post-op) in cortisol, IL1 and IL6 will be calculated together with their standard deviations.

SECONDARY OUTCOMES:
The area under the curve for insulin concentration.
Maximum change in IL2, IL3, IL8 and IL10 from baseline to day 3 post-op.
Description of other blood parameters related to stress response.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Craig Carr, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom